CLINICAL TRIAL: NCT01135953
Title: Investigating Methods to Enhance the Excitatory Effects of Transcranial Direct Stimulation (tDCS)
Brief Title: Methods to Enhance Transcranial Direct Stimulation (tDCS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Associate Professor Colleen Loo, School of Psychiatry, University of New South Wales
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: HREC09344
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Healthy Volunteers; Brain Excitation
Keywords: Brain excitation; transcranial Direct Stimulation; administration pattern
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Cycloserine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ARM 1 - CONTROL (Experimental): Subject given tDCS every day of the week (5 sessions) at 2 mA.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Arm 2 - INCREASING (Experimental): Subjects given increasing intensity during tDCS across the week (Monday 1mA, Tuesday 1.5mA, Wednesday 1.5 mA, Thursday 2 mA, Friday 2mA).
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- ARM 3 - CYCLOSERINE (Experimental): D-cycloserine (100 mg) given on the Monday and Thursday sessions, administering tDCS at 2 mA.
  Interventions: Other: Transcranial direct Stimulation (tDCS) and D-cycloserine

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS applied to to motor cortex every weekday (5 sessions), at 2mA ,during 20 minutes.Conductive rubber electrodes (7 x 5 cm = 35 cm2) covered by sponges soaked in saline will be used, held in place by a band. The current will be gradually increased to the level of 2 mA over 30 seconds (to avoid the sensation of a flash).
  Other Names: tDCS (Eldith DC-Stimulator (CE certified)
  Arms: ARM 1 - CONTROL
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS applied to the motor cortex every day of the week during 20 minutes, at 1mA first session, 1.5 mA second and third sessions, and 2mA fourth and fifth sessions, during 20 minutes. Conductive rubber electrodes (7 x 5 cm = 35 cm2) covered by sponges soaked in saline will be used, held in place by a band. The current will be gradually increased over 30 seconds (to avoid the sensation of a flash).
  Other Names: Eldith DC-Stimulator (CE certified)
  Arms: Arm 2 - INCREASING
Other: Transcranial direct Stimulation (tDCS) and D-cycloserine — Transcranial Direct Stimulation applied to the motor cortex every day of the week (5 sessions) at 2mA, during 20 minutes. Conductive rubber electrodes (7 x 5 cm = 35 cm2) covered by sponges soaked in saline will be used, held in place by a band. The current will be gradually increased to the level of 2 mA over 30 seconds (to avoid the sensation of a flash).
  D-cycloserine, administered orally (capsules), 100 mg, twice a week (Monday and Thursday), prior to the tDCS session.
  Other Names: tDCS - Eldith DC-Stimulator (CE certified); D-cycloserine, Seromycin Pulvules, 100 mg
  Arms: ARM 3 - CYCLOSERINE

SUMMARY:
tDCS has been shown to be an effective treatment for depression. However, tDCS is a relatively new clinical tool and more needs to be understood about its use. This study hopes to further the field of knowledge by examining how tDCS should be optimally used. Application of tDCS in clinical trials of depression is typically to the prefrontal cortex, but in this project, tDCS application will be to the motor cortex as it provides a more ready measure of excitability. Excitability will be measured using Transcranial Magnetic Stimulation (TMS) to the motor cortex and electromyography (EMG) recordings from peripheral muscles stimulated. Using a cross-over three-arm design this study aims to investigate whether daily tDCS administered in increasing intensity across sessions leads to greater and lasting effects on brain excitability than keeping the intensity at a same dose across the days and whether the excitatory effect could be enhanced with D-cycloserine, a medication known to prolong the excitatory effects of a single session of tDCS. This in turn will inform on how to optimize tDCS for therapeutic applications, e.g treatment of depression. The study hypothesis is that 5 sessions of tDCS with a dose of D-cycloserine given on the Monday and Thursday sessions will result in more sustained effect on motor cortex excitability than 5 sessions of tDCS alone. The second hypothesis is that the gradational increases in tDCS intensity over 5 sessions will result in greater motor cortex excitability than 5 sessions of tDCS where intensity is kept constant across sessions.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Right handed (> 18/20 on the Edinburgh Handedness)
* Aged 18-40

Exclusion Criteria:

* Mental illness
* General medical illness
* Neurological illness, epilepsy
* Alcohol use above National Health and Medical Research Council (NHMRC) guidelines
* Smokers
* Excessive caffeine intake
* Illicit drug use
* Herbal medication use
* Electronic implant, e.g, cochlear implant, pacemaker
* Musculoskeletal problem in the arm

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in brain excitability measured through motor evoked potentials (MEP) 0 to 120 minutes after tDCS session. | Pre-treatment, post treatment at minute 0, minute 5, minute 10, minute 15, minute 20, minute 25, minute 30, minute 60, minute 90, minute 120.

CONTACTS AND LOCATIONS:
Locations (1):
- Black Dog Institute, University of New South Wales, Sydney, New South Wales, Australia

REFERENCES:
- See also: Black Dog Institute website — http://www.blackdoginstitute.org.au